CLINICAL TRIAL: NCT03756311
Title: Expanded Access to NanoPac
Status: No longer available | Type: Expanded Access
Sponsor: NanOlogy, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: NANOPAC-EA
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Pancreatic Carcinoma; Prostate Cancer; Lung Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Lung Neoplasms | interventions — Powders; Suspensions; Paclitaxel

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: NanoPac (sterile nanoparticulate paclitaxel) Powder for Suspension
  Other Names: Paclitaxel

SUMMARY:
NanOlogy may consider offering expanded access to NanoPac for patients who do not meet the enrollment criteria of clinical trials in progress.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult